CLINICAL TRIAL: NCT03792373
Title: Effects of Frailty on Outcomes After Elective Noncardiac Surgery -a Prospective Cohort Study
Brief Title: Hospital Ederly Life Program for Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Jian-jun Yang, Principal Investigator, Zhongda Hospital
Other Study IDs: HELP
Record Dates: First submitted 2018-12-25; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: To Investigate the Mortality of the Frailty Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- frailty
- nonfrailty

SUMMARY:
Frailty is the clinically recognizable medical condition, also called syndrome or phenotype, that is, the result of processes leading to an increased vulnerability for serious deteriorations in health and the diminished ability to cope with physical stressors. Recently, frailty has emerged as a significant risk factor for adverse postoperative outcomes. It is related to declines in energy, strength, and function as well as to an increased inflammatory state, including elevated levels of interleukin 6 (IL-6), C-reactive protein (CRP), and anelevated white blood cell count . Frailty, as defined Frailty, as defined in the landmark paper by Fried, included at least three of five of the following criteria: unintentional loss of weight, low physical activity, low energy, low grip strength, and a slowed walking speed. Since then, various frailty scoring lists have been designed to optimize the predictive value. One of these is the Edmonton Frail Scale (EFS), an instrument that can be assessed quickly, using only a simple questionnaire which usually does not require more than five minutes to be completed and which covers most domains of functioning, making it easy and fast to get a reliable impression of the degree of frailty.The aim of this study was to determine which factors,with emphasis on frailty, significantly influence postoperative outcome after elective noncardiac surgery as measured by the Comprehensive Complication Index (CCI).

ELIGIBILITY:
Inclusion Criteria:

* elective noncardiac surgery

Exclusion Criteria:

* patients who don't cooperate

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: ≥65 years
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
one-year mortality | 2019.02-2020.02
  To investigate the one-year mortality of the frailty patients

CONTACTS AND LOCATIONS:
Overall Officials: Gaojun Teng, PhD, Study Chair — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mao M, Wang LY, Zhu LY, Wang F, Ding Y, Tong JH, Sun J, Sun Q, Ji MH. Higher serum PGE2 is a predicative biomarker for postoperative delirium following elective orthopedic surgery in elderly patients. BMC Geriatr. 2022 Aug 19;22(1):685. doi: 10.1186/s12877-022-03367-y. PMID 35982410